CLINICAL TRIAL: NCT01683877
Title: PROSPECTIVE RANDOMIZED CONPARISON OF ELECTRONIC DIATHERMY VERSUS FLOSEAL IN HEMOSTASIS AFTER LAPAROSCOPIC OVARIAN CYSTECTOMY
Brief Title: Efficacy Study of FloSeal in Hemostasis After Laparoscopic Ovarian Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FloSeal-OC
Record Dates: First submitted 2012-09-03; First posted 2012-09-12 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Benign Ovarian Tumor
MeSH Terms: interventions — Electrocoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FloSeal group (Experimental): After laparoscopic ovarian cystectomy, hemostasis will be performed using FloSeal (1 vial of FloSeal 5mL per unilateral ovarian cystectomy)
  Interventions: Procedure: FloSeal application
- Electrocautery group (Active Comparator): After laparoscopic ovarian cystectomy, hemostasis will be performed using electrocautery
  Interventions: Procedure: Electrocautery

INTERVENTIONS:
Procedure: FloSeal application — After laparoscopic ovarian cystectomy, hemostasis will be performed using FloSeal (1 vial of FloSeal 5mL per unilateral ovarian cystectomy)
  Arms: FloSeal group
Procedure: Electrocautery — After laparoscopic ovarian cystectomy, hemostasis will be performed using electrocautery
  Arms: Electrocautery group

SUMMARY:
To compare the efficacy in postoperative hemostasis and in sparing postoperative ovarian function between FloSeal and Electrocauterization in laparoscopic ovarian cystectomy

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* Patients who is planned to undergo laparoscopic ovarian cystectomy
* American Society of Anesthesiologists Physical Status classification (ASA PS) 1-2
* Patients with adequate bone marrow, renal and hepatic function:

WBC > 3,000 cells/mcl Platelets >100,000/mcl Creatinine <2.0 mg/dL Bilirubin <1.5 x normal and SGOT or SGPT <3 x normal

* Patient must be suitable candidates for surgery
* Patients who have signed an approved Informed Consent

Exclusion Criteria:

* Patients with a history of pelvic or abdominal radiotherapy;
* Patients who are pregnant or nursing
* Patients who is receiving or requires hormone replacement therapy after surgery
* Patients who is undergoing hysterectomy at this time
* Patients who is undergoing unilateral or bilateral oophorectomy
* Previous history of ovarian cystectomy or oophorectomy
* Patients with contraindications to surgery
* Unfit for Surgery: serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Patient compliance and geographic proximity that do not allow adequate follow-up.
* Hormone therapy within 3 months before surgery

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hemostasis time | Immediately after operation

SECONDARY OUTCOMES:
Ovarian function after surgery | within 6 months after surgery
Operative time | 1 day (Immediately after surgery)
Intraoperative blood loss | During surgery
Postoperative drainage duration | within 1 week after surgery
Length of postoperative stay | within 1 month after surgery
Postoperative complications | within 1 months after surgery
  Postoperative complications will be evaluated with Dindo's classification for postoperative complication and CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hyun Nam, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea